CLINICAL TRIAL: NCT04427202
Title: Ending Transmission of HIV, HCV, and STDs and Overdose in Rural Communities of People Who Inject Drugs (ETHIC)
Acronym: ETHIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Southern Illinois University (Other); Community Action Place, Inc. (Other); New York University (Other); University of Illinois at Chicago (Other); University of Washington (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB17-1630; 4UH3DA044829-03 (NIH)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-08

CONDITIONS: HIV; Hepatitis C; Opioid-use Disorder; Injection Drug Use
Keywords: HIV; Hepatitis C; Opioid-use Disorder; Injection Drug Use; Harm Reduction Services
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Referral to harm reduction services (Other): Participants will be taken through the study survey and interview, blood and urine toxicology testing and given a referral to a harm reduction organization.
  Interventions: Behavioral: Referral to harm reduction services

INTERVENTIONS:
Behavioral: Referral to harm reduction services — Participants are referred to harm reduction services

SUMMARY:
This study will evaluate the referral to harm reduction services (HRS) including syringe services, naloxone overdose prevention, substance use treatment referral, HIV, HCV, and STD testing and referral and linkage to care through capacity building of existing programs through client services data.

DETAILED DESCRIPTION:
This is a prospective longitudinal Type 1 Hybrid Implementation Effectiveness Study on the expansion of harm reduction services for people who inject drugs (PWID) and people who use opioids (PWUO) residing in high risk areas of rural southern Illinois. This study record describes one component of the larger Ending transmission of HIV, HCV, and STDs and overdose in rural communities of people who inject drugs (ETHIC) study Community Response Plan (CRP) framework, specifically the expansion of harm reduction services intervention (HRS). The aim is to assess the effectiveness of expansion of evidenced based harm reduction services through our CRP framework comprising: a) geographically targeted recruitment based on hot spot and vulnerability analyses, b) community engagement, c) recruitment via Respondent Driven Sampling (RDS), d) expanded surveillance for HIV and HCV, and e) concomitant HCV and opioid use treatment capacity expansion through the Extension of Community Healthcare Outcomes (ECHO) model. Examination of facilitators and barriers impacting implementation of service delivery is evaluated through mixed methods process evaluation. The Type 1 Hybrid design is supported by conditions including the existing evidence based for benefits and minimal harm of "harm reduction services" and strong base for applicability of this intervention in the study setting (ie rural opioid use)

ELIGIBILITY:
Inclusion Criteria:

* 15 years of age and older
* Injected any drug in the past 30 days
* Used any opioids non-medically in the past 30 days
* English speaking
* Able to provide informed consent at the time of the study visit

Exclusion Criteria:

* Less than 15 years of age
* Not injected any drug in the past 30 days
* Not used any opioids non-medically in past 30 days
* Non-English speaking
* Has not injected any opioid drug to get high in the past 30 days
* Unable to provide informed consent at the time of the study visit

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mai Pho, PhD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Southern Illinois University, Carbondale, Illinois
  - The Community Action Place, Inc., Murphysboro, Illinois

IPD SHARING:
Plan to Share IPD: Yes
The ETHIC study is participating site of the Rural Opioid Initiative (ROI), a collaborative funded by NIDA. The ROI includes a Data Coordinating Center (DCC) housed at the University of Washington. The University of Chicago will submit de-identified data from the study to the DCC as covered under a data use agreement for the purposes of performing cross-site analyses using a harmonized data set. No parties outside of the ROI will have access to the combined dataset. All project proposals will be subject to approval by the ROI. The data will be available after encrypted submission to the DCC and will remain for the duration in accordance to the data use agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available at the DCC for the time frame indicated in the data use agreement.
Access Criteria: Data will be shared among researchers in the Rural Opioid Initiative (ROI) cooperative agreement as described above

REFERENCES:
- [Derived] Rains A, York M, Bolinski R, Ezell J, Ouellet LJ, Jenkins WD, Pho MT. Attitudes toward harm reduction and low-threshold healthcare during the COVID-19 pandemic: qualitative interviews with people who use drugs in rural southern Illinois. Harm Reduct J. 2022 Nov 19;19(1):128. doi: 10.1186/s12954-022-00710-9. PMID 36403075
- [Derived] Walters SM, Bolinski RS, Almirol E, Grundy S, Fletcher S, Schneider J, Friedman SR, Ouellet LJ, Ompad DC, Jenkins W, Pho MT. Structural and community changes during COVID-19 and their effects on overdose precursors among rural people who use drugs: a mixed-methods analysis. Addict Sci Clin Pract. 2022 Apr 25;17(1):24. doi: 10.1186/s13722-022-00303-8. PMID 35468860

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort: Participants will be taken through the study survey and interview, blood and urine toxicology testing and given a referral to a harm reduction organization.
Period: Baseline
Arm/Group | Cohort
Started | 306
Completed | 306
Not Completed | 0
Period: 6 Months
Arm/Group | Cohort
Started | 306
Completed | 74
Not Completed | 232
Period: 12 Months
Arm/Group | Cohort
Started | 74
Completed | 44
Not Completed | 30
Period: 18 Months
Arm/Group | Cohort
Started | 44
Completed | 17
Not Completed | 27
Period: 24 Months
Arm/Group | Cohort
Started | 17
Completed | 4
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: Participants who consented and completed the baseline survey.
Arm/Group | Cohort
Number analyzed (Participants) | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 297
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 199
  Sex: Female | 106
  Sex: Intersex | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 296
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 63
  White | 230
  More than one race | 7
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Participants Who Received Referrals to the Harm Reduction Services Organization
Description: Number of participants who accept referral to the intervention (divided by the total enrolled who did not have previous engagement prior to the study with the harm reduction services organization).
Time Frame: 2 years
Population: These participants who did not have previous engagement prior to the study with the harm reduction services organization.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort: Participants who have not previous engaged at the HRSO
Arm/Group | Cohort
Number analyzed (Participants) | 207
Participants | 121

2. Secondary Outcome: Number of Locations Where Participants Received Most of Syringes or Needles
Description: Number of unique zip codes that participants received most of their syringes or needles based on mobile unit delivery.
Time Frame: 2 years
Measure: Number; unit: Unique zip codes
Groups:
- Cohort: Total participants who responded at baseline up to 24 months.
Arm/Group | Cohort
Number analyzed (Participants) | 306
Unique zip codes | 92

3. Secondary Outcome: Number of Times Sterile Syringes and/or Equipment Obtained From an Intervention
Description: This was counted as the number of visits made by the hard reduction service organization to distribute sterile syringes and/or equipment.
Time Frame: 2 years
Measure: Mean (Full Range); unit: Visits
Arm/Group | Cohort
Number analyzed (Participants) | 306
Visits | 2.5 [0 to 30]

4. Secondary Outcome: Number of Times Participants Used a Syringe or Needle That They Knew Was Used by Somebody Else
Description: "How many times (encounters) in the past 30 days did you inject using a syringe or needle that you know had been used by somebody else?"
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Encounters
Arm/Group | Cohort
Number analyzed (Participants) | 306
Encounters | 0.9 (3.0)

5. Secondary Outcome: Number of Times Participants Used a Cotton, Cooker, Spoon, or Water for Rinsing or Mixing That They Knew Was Used by Somebody Else
Description: "How many times (encounters) in the past 30 days did you use a cotton, cooker, spoon or water for rinsing or mixing that you know had been used by somebody else?"
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Encounters
Arm/Group | Cohort
Number analyzed (Participants) | 306
Encounters | 2.5 (9.5)

6. Secondary Outcome: Number of Times Participants Let Someone Else Use a Cotton, Cooker, Spoon, or Water for Rinsing or Mixing After They Used it
Description: "How many times (encounters) in the past 30 days did you let someone else use a cotton, cooker, spoon, or water for rinsing or mixing after you used it?"
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Encounters
Arm/Group | Cohort
Number analyzed (Participants) | 306
Encounters | 2.3 (8.4)

7. Secondary Outcome: Number of Participants With Drive Time Less Than 30 Minutes to Nearest Syringe or Needle Exchange
Description: Number of participants with drive time less than 30 minutes to nearest syringe or needle exchange.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 306
Participants | 148

8. Secondary Outcome: Number of Participants That Currently Have Naloxone
Description: "Do you currently have naloxone or Narcan with you or at home?"
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 306
Participants | 93

9. Secondary Outcome: Number of Participants Who Received Substance Use Disorders (SUD) Treatment Referrals
Description: Total number of participants who received a substance use disorder referrals made by the hard reduction services organization.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 306
Participants | 102

10. Secondary Outcome: Total Number of Participants Who Received an HIV Screening
Description: Total number of tests that participants screened for HIV, from baseline to follow-up.
Time Frame: 2 years
Population: Participants who already knew their HIV+ diagnoses prior to this study (n=4) and thus, removed from the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 302
Participants | 288

11. Secondary Outcome: Total Number of Participants Who Received an HCV Screening
Description: Total participants screened for HCV at least once during baseline and follow-up. For those who had a HCV reactive test were then later referred to further services.
Time Frame: 2 years
Population: Participants who already were told they had HCV prior to this study (n=76) were removed from the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 230
Participants | 213

12. Secondary Outcome: Number of Participants With Knowledge of PrEP
Description: "Have you ever heard of medicine people can take to prevent HIV?"
Time Frame: 6 months
Population: Participants did not respond to question (n=5)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort: Total participants who responded at baseline up to 6 months.
Arm/Group | Cohort
Number analyzed (Participants) | 301
Participants | 155

13. Secondary Outcome: Number of Participants Diagnosed With HIV Who Have Access to HIV Care
Description: Total number of participants who were newly diagnosed with HIV during the study period.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 306
Participants | 0

14. Secondary Outcome: Number of Participants Diagnosed With HCV Who Have Access to HCV Care
Description: Total number of participants who were newly diagnosed with chronic Hep C who were referred to Hep C care.
Time Frame: 2 years
Population: Total number of participants who had a positive confirmatory HCV test (e.g. positive viral load).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort
Number analyzed (Participants) | 11
Participants | 11

15. Secondary Outcome: Number of Times a Participant Engaged in Condomless Sex (Vaginal or Anal)
Description: "In the last 30 days, how many times did you have vaginal or anal sex without a condom?"
Time Frame: 6 months
Population: A number of participants did not respond to this question (n=10).
Measure: Mean (Standard Deviation); unit: Encounters
Arm/Group | Cohort
Number analyzed (Participants) | 296
Encounters | 9.9 (16.2)

ADVERSE EVENTS:
Time Frame: Study period from baseline to 24-month follow-up.
Arm/Group | Cohort
All-Cause Mortality (participants affected / at risk) | 4/306
Serious Adverse Events (participants affected / at risk) | 5/306
Other Adverse Events (participants affected / at risk) | 0/306
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort (N=306)
Deaths (General disorders) | 4 (4) — Overdose death
Suicidial Ideation (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT04427202/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT04427202/SAP_001.pdf